CLINICAL TRIAL: NCT05101616
Title: A Pilot Study of Neoadjuvant Chemotherapy With or Without Camrelizumab for Locally Advanced Gastric Cancer: a Single-center, Open-label, Randomized Controlled Trial
Brief Title: A Pilot Study of Neoadjuvant Chemotherapy With or Without Camrelizumab for Locally Advanced Gastric Cancer
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: difficult in enrolling participants
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Camrelizumab-GC-neoadjuvant
Record Dates: First submitted 2021-10-28; First posted 2021-11-01 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; neoadjuvant chemotherapy; immunotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- camrelizumab+chemotherapy (Experimental): neoadjuvant treatment with camrelizumab+chemotherapy
  Interventions: Drug: camrelizumab+chemotherapy
- chemotherapy (Active Comparator): neoadjuvant treatment with chemotherapy
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: camrelizumab+chemotherapy — camrelizumab 200mg，ivdrip，q3w； albumin nanoparticle of paclitaxel 260 mg/m2、 ivdrip，d1，q3w； oxaliplatine 85mg/m2、ivdrip，d1，q3w； S-1 40 mg/m2，po, bid，d1~d14，q3w. 3 cycles.
  Arms: camrelizumab+chemotherapy
Drug: Chemotherapy — albumin nanoparticle of paclitaxel 260 mg/m2、 ivdrip，d1，q3w； oxaliplatine 85mg/m2、ivdrip，d1，q3w； S-1 40 mg/m2，po, bid，d1~d14，q3w. 3 cycles.
  Arms: chemotherapy

SUMMARY:
It is a single-center, open-lable, randomized controlled trial to prospectively investigate the effectiveness and safety of Camrelizumab combined with DOS regimen chemotherapy in neoadjuvant treatment of patients with locally advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily join the study and sign an informed consent form, have good compliance and cooperate with follow-up;
2. Male or female patients between the ages of 18-75;
3. Patients diagnosed as gastric adenocarcinoma by histology or cytology;
4. Stage: Locally advanced stage (T3-4aN1-3M0);
5. Have not received other immunotherapy drugs or chemotherapy drugs in the past;
6. ECOG (Eastern US Cooperative Oncology Group) score: 0-1 points;
7. Has sufficient organ and bone marrow function

Exclusion Criteria:

1. Other malignant tumors that have appeared or are currently suffering from within 5 years, except for cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) ) And T1 (tumor infiltration basement membrane)];
2. A distant metastasis occurs;
3. Those who have multiple factors that affect oral medications (such as inability to swallow, chronic diarrhea, etc.);
4. Accompanied by pleural effusion or ascites, causing respiratory syndrome (NCI-CTC AE V5.0 grade ≥ 2 dyspnea);
5. Patients with any severe and/or uncontrollable disease；
6. Patients with gastrointestinal diseases with bleeding tendency (such as active gastrointestinal ulcers) or patients determined by the researcher to cause gastrointestinal bleeding, perforation or obstruction
7. Patients whose imaging shows that the tumor has invaded the tissues around important blood vessels or the investigator judges that the tumor is likely to invade important blood vessels and cause fatal bleeding during the follow-up study;
8. Received glucocorticosteroid or immunosuppressive therapy within 7 days before grouping;
9. Regardless of the severity, patients with any signs of bleeding or medical history; within 4 weeks before grouping, patients with any bleeding or bleeding events NCI-CTC AE V5.0 grade ≥ 3, unhealed wounds, ulcers Or fracture
10. Those who have had arterial/venous thrombotic events within 6 months, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis and pulmonary embolism;
11. People with a history of psychotropic drug abuse and unable to quit or have mental disorders;
12. Participated in other anti-tumor drug clinical trials within four weeks;
13. According to the judgment of the investigator, those with concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study;
14. Female patients who are pregnant or breastfeeding;
15. Known hypersensitivity to any study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
major pathologic response rate | one month after surgery
  complete or subtotal regression (<10% residual tumor per tumor bed)

SECONDARY OUTCOMES:
complete pathologic response rate | one month after surgery
  complete regression (no residual tumor per tumor bed)
R0 resection rate | one month after surgery
  surgically removed tissue without residual cancer cells
Overall survival | 3 years
  the time from the start of randomization to death due to any cause.
Disease-free survival | 3 years
  the time from the start of randomization to the incurable resection, local recurrence or metastasis, or death from any cause.
perioperative complications | the time from the start of randomization to 3 months after surgery
  perioperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China